CLINICAL TRIAL: NCT05281081
Title: Comparison of Intra-Peritoneal Instillation of Levobupivacaine With Morphine Hydrochloride Versus Levobupivacaine With Magnesium Sulfate for Post-Operative Pain Relief After Laparoscopic Cholecystectomy
Brief Title: Intraperitoneal Instillation of Levobupivacaine With Morphine Versus Levobupivacaine With Magnesium Sulfate for Postoperative Analgesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Islam Mokhtar Ahmed, lecturer of anesthesia and intensive care, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Soh-Med-22-02-27
Record Dates: First submitted 2022-03-06; First posted 2022-03-15 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- levobupivacaine with morphine (Active Comparator): 30 patients will have intraperitoneal instillation of levobupivacaine with added morphine at the end of laparoscopic cholecystectomy operation
  Interventions: Drug: intraperitoneal levobupivacaine and morphine
- levobupivacaine with magnesium sulfate (Experimental): 30 patients will have intraperitoneal instillation of levobupivacaine with added magnesium sulfate at the end of laparoscopic cholecystectomy operation
  Interventions: Drug: intraperitoneal levobupivacaine and morphine

INTERVENTIONS:
Drug: intraperitoneal levobupivacaine and morphine — istillation of the peritoneum with levobupivacaine mixture with morphine

SUMMARY:
This is a prospective randomized study that included 60 patients and was divided into two equal groups of patients who were scheduled for LC, Ages 18 and 60 years, both sexes, ASA I-II and BMI 19 - 39. Group A received 30 ml levobupivacaine (0.25%) plus 3 mg morphine intraperitoneal at the site of surgery in the bed of the gallbladder via the navel port with the patient in a Trendelenburg position, Group B received 30 ml levobupivacaine (0.25%) plus 50 mg/kg magnesium sulfate in the same pattern as in the A group.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were scheduled for L.C,
* Ages 18 and 60 years
* ASA I-II and
* BMI 19 - 39

Exclusion Criteria:

* Patients with hepatic or renal dysfunction
* use of opioids 24 hrs prior to the study
* treatment with steroids prior to surgery
* drug or alcohol abuse, allergy to any of the study drugs
* chronic pain syndrome as a result of neurological disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
reduction of postoperative pain | 8 hours
  reduction of post operative visual analogue score

CONTACTS AND LOCATIONS:
Locations (1):
- ‪Khalid abdelal‬, Sohag, Egypt